CLINICAL TRIAL: NCT00254319
Title: Phase II Trial of Bevacizumab (Avastin) Plus Pemetrexed (Alimta) and Carboplatin in Previously Untreated Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Previously Untreated Advanced Non-Small Cell Lung Cancer (NSCLC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Cooper Health System (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVF3158'S
Record Dates: First submitted 2005-11-14; First posted 2005-11-16 (Estimated); Last update posted 2005-11-16 (Estimated); Status verified 2005-11

CONDITIONS: Untreated Advanced Non-Small Cell Lung Cancer
MeSH Terms: interventions — Bevacizumab; Pemetrexed

INTERVENTIONS:
Drug: Avastin, Alimta

SUMMARY:
Avastin is a novel antiangiogenic agent that has recently been shown to improve response rates and survival of patients with advanced nonsquamous non-small cell lung cancer when added to front-line carboplatin/paclitaxel chemotherapy, and is now being routinely incorporated into the treatment of these patients. Alimta is a recently approved chemotherapeutic that has shown activity against non-small cell lung cancer when given alone and in combination with carboplatin, has a favorable toxicity profile andrequires only a brief (10 minute) infusion time. Therefore we propose to study the combination of Avasin, Alimta, and Carboplatin administered as front-line therapy to patients with advanced nonsquamous non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

I am 18 years of age or older. I have advanced non-small lung cancer. I have not had any major surgical procedures within 28 days prior to my starting treatment.

I have high blood pressure that is controlled. I am not on heparin, coumadin or lovonox for treatment of medical conditions. I do not have serious wound healing problems. I have not received any previous treatment, except radiation therapy for my disease.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: James Stevenson, M.D., Principal Investigator — The Cooper Health System
Locations (1):
- The CINJ at Cooper University Hospital, Voorhees Township, New Jersey, United States